CLINICAL TRIAL: NCT05826015
Title: Phase I/IB of AVB-500 (Batiraxcept) in Combination With Paclitaxel in Recurrent High Grade Uterine Cancer
Brief Title: AVB-500 (Batiraxcept) in Combination With Paclitaxel in Recurrent High Grade Uterine Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Trial did not go forward
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Aravive, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202306082
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Recurrent High Grade Uterine Cancer
Keywords: Batiraxcept; AVB-500; uterine serous; high-grade endometrioid; paclitaxel
MeSH Terms: interventions — Paclitaxel; AVB-500 fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Paclitaxel + AVB-500 (Experimental): Patients will receive up to 9 21-day cycles of paclitaxel + AVB-500. Patients will receive AVB-500 via intravenous (IV) infusion at the assigned dose level on days 1, 8, and 15 of each cycle. Patients will receive IV paclitaxel at a dose of 175 mg/m^2 on day 1 of each cycle. After 3 cycles, patients will be assessed for disease response. Patients who have progression will not continue on treatment. Patients who have a partial response or stable disease will continue on treatment for another 3 cycles of paclitaxel + AVB-500 at the assigned dose. Patients will be assessed for response again at the end of 6 cycles and may continue on treatment if they have partial response (PR) or stable disease (SD). Up to 9 cycles of treatment with paclitaxel + AVB-500 may be given. At the end of the 9 cycles, patients with a SD or PR can continue on maintenance AVB-500 until progression. Patients with complete response will continue single agent AVB-500 as maintenance therapy until progression.
  Interventions: Drug: Paclitaxel; Drug: Batiraxcept

INTERVENTIONS:
Drug: Paclitaxel — IV over 3 hours
  Other Names: Taxol
Drug: Batiraxcept — IV over 60 minutes
  Other Names: AVB-500

SUMMARY:
The purpose of this study is to determine safety and tolerability of AVB-500 when given in combination with paclitaxel in patients with recurrent high-grade uterine cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent, FIGO grade 3 endometrioid, serous, or mixed high grade uterine or endometrial cancer. Patients must have experienced either prior progression on a platinum-based therapy or intolerance to platinum. Patients with dMMR or MSI-H tumors or targetable HER2 alterations are required to have received prior therapy with appropriate targeted agents.
* Patients must have disease that cannot be managed by local therapy.
* Measurable disease by RECIST 1.1
* Women or transgender men with a uterus who are at least 18 years of age.
* ECOG performance status ≤ 2
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1.5 K/cumm
  * Platelets ≥ 100 K/cumm
  * Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN (unless liver metastases are present in which case AST/ALT must be ≤ 5.0 x IULN)
  * Serum creatinine < 2.0 mg/dL or < 177 µmol/L OR calculated or measured creatinine clearance ≥ 40 mL/min (using Cockcroft-Gault equation)
  * INR ≤ 1.5 x IULN
  * aPTT ≤ 1.5 x IULN
* The effects of AVB-500 on the developing human fetus are unknown. For this reason and because chemotherapeutic agents are known to be teratogenic, patients of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a patient become pregnant or suspect pregnancy while participating in this study, the treating physician must be informed immediately.
* Subjects who have received prior treatment with trastuzumab, pembrolizumab, or dostarlimab can enroll in the study.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Any prior treatment with AVB-500
* A history of other malignancy with the exception of malignancies for which all treatment was completed at least 2 years before registration and the patient has no evidence of disease.
* Currently receiving any other (non-study) cytotoxic chemotherapy, radiation, targeted treatment, or immunotherapy within 4 weeks prior of start of study treatment.
* Currently receiving any other investigational agents or has received an investigational agent within 4 weeks of start of study treatment.
* Known brain metastases. Patients with known brain metastases must be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to AVB-500 or other agents used in the study.
* Abnormal gastrointestinal function, defined as Grade >2 diarrhea, constipation, nausea, vomiting, or abdominal pain. This includes GI obstruction or bleeding or signs/symptoms thereof within 3 months of study enrollment. Patients with a history of abdominal fistula will be considered eligible if the fistula was surgically repaired or has healed, there has been no evidence of fistula for at least 6 months, and patient is deemed to be at low risk of recurrent fistula.
* Significant cardiac disease history including:

  * Clinically significant atrial or ventricular arrhythmias requiring treatment
  * Medically controlled congestive heart failure
  * Significant angina or clinically and/or electrocardiographically documented myocardial infarction within the past year
  * Clinically significant valvular disease
* Non-healing wound, ulcer, or bone fracture.
* Known active hepatitis; ongoing systemic bacterial, fungal, or viral infection.
* History or evidence upon physical examination of CNS disease, including primary brain tumor, seizures not controlled with standard medical therapy, or history of CVA, TIA, or subarachnoid hemorrhage within 6 months of the first date of treatment on this study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* History of major surgical procedure within 14 days prior to start of study treatment.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended. Recommend exclusion of specific ART agents based on predicted drug-drug interactions (i.e. for sensitive CYP3A4 substrates, concurrent strong CYP3A4 inhibitors (ritonavir and cobicistat) or inducers (efavirenz) should be contraindicated).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-31 (Estimated); Primary Completion 2029-06-03 (Estimated); Study Completion 2034-06-04 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of treatment-emergent adverse events | From start of treatment though 30 days after the last dose of AVB-500 (estimated to be 31 weeks)
  -Graded by CTCAE v.5.

SECONDARY OUTCOMES:
Serum sAXL and GAS6 ratio | At baseline
Pharmacokinetic (PK) parameters (including Cmax) as determined from AVB-500 serum levels | Cycle 1 Day 1 pre-infusion, Cycle 1 Day 1 post-infusion, Cycle 1 Day 15 pre-infusion, and subsequent cycles day 1 pre-infusions (each cycle is 21 days)
Pharmacokinetic (PK) parameters (including Tmax) as determined from AVB-500 serum levels | Cycle 1 Day 1 pre-infusion, Cycle 1 Day 1 post-infusion, Cycle 1 Day 15 pre-infusion, and subsequent cycles day 1 pre-infusions (each cycle is 21 days)
Pharmacodynamic effects as determined by changes from baseline in serum GAS6 levels | Cycle 1 Day 1 pre-infusion, Cycle 1 Day 1 post-infusion, Cycle 1 Day 15 pre-infusion, and subsequent cycles day 1 pre-infusions (each cycle is 21 days)
Overall response rate (ORR) | Through completion of treatment (estimated to be 27 weeks)
  -Defined as the proportion of subjects who have a partial or complete response to therapy
Progression-free survival (PFS) | Through completion of follow-up (estimated to be 5 years and 27 weeks)
  -Defined as the time from start of treatment to the first radiologically documented disease progression, or death, whichever comes first. The alive patients without radiologically documented disease progression are censored at the last follow-up.
Recommended Phase 2 dose (RP2D) of AVB-500 in combination with paclitaxel | Through completion of cycle 1 (cycle=21 days) for all patients (estimated to be 48 months and 3 weeks)
Incidence of anti-drug antibodies (ADA) | Day 1 of each cycle (cycle-21 days) and end of treatment (estimated to be 27 weeks)
Overall survival (OS) | Through completion of follow-up (estimated to be 5 years and 27 weeks)
  -Defined as the time from start of treatment to death. The alive patients are censored at the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: David G Mutch, M.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu